CLINICAL TRIAL: NCT04942665
Title: Low Dose ICG for Near-infrared Fluorescence Imaging of Biliary Tract and Tumors
Brief Title: Low Dose ICG for Biliary Tract and Tumor Imaging
Acronym: ICG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Society of University Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB202100388; OCR40380 (Other: UF OnCore); PRO00043219 (Other: UFIRST)
Record Dates: First submitted 2021-05-28; First posted 2021-06-28 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Cholecystitis; Hepatocellular Carcinoma; Liver Metastases
Keywords: Biliary Tract; Indocyanine Green (ICG); Tumors; Near-infrared Fluorescence
MeSH Terms: conditions — Cholecystitis; Carcinoma, Hepatocellular; Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Adult patients scheduled to undergo a laparoscopic hepatic or biliary operation will be randomized to two groups 1) low dose (0.05 mg) or 2) standard dose (2.5 mg) of ICG preoperatively on the day of surgery. Patients with a history of adverse reactions or known allergy to ICG, iodine, or iodine dyes will be excluded.
Who Masked: Participant, Investigator
Masking Description: To mask the investigator randomization will be done with envelopes for this study and the dose given to the patient prior to surgery with the investigator not being aware of the amount given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Low Dose (Experimental): Prior to surgery these patients will be given a ICG dose of 0.05 mg IV.
  Interventions: Drug: Indocyanine green; Device: PINPOINT Endoscopic Fluorescence
- Standard Dose (Placebo Comparator): Prior to surgery these patients will be given the ICG standard dose of 2.5 mg IV.
  Interventions: Drug: Indocyanine green; Device: PINPOINT Endoscopic Fluorescence

INTERVENTIONS:
Drug: Indocyanine green — Low dose or standard dose ICG will be administered by the anesthesiologist as guided by the study coordinator at the beginning of the case, at two points during the operation (1- prior to the dissection of the biliary tract and 2- upon completion of the dissection and establishment of the critical view of safety).
  Other Names: ICG
Device: PINPOINT Endoscopic Fluorescence — The PINPOINT Endoscopic Fluorescence Imaging System (Stryker Corporation, Kalamazoo, Michigan) will be used. This device enables the surgeon to simultaneously see real-time, high-definition visible-range and NIR fluorescence videos and to superimpose them. It is currently approved by the FDA for intraoperative near-infrared fluorescence imaging.
  Other Names: NIRF

SUMMARY:
Near-infrared fluorescence (NIRF) imaging after an intravenous injection of indocyanine green (ICG) allows for the intraoperative identification of liver anatomy. The investigators have new data that a much lower dose improves this visualization. Confirmation of this hypothesis would mean that ICG can be administered on the same day of surgery in order to augment real-time intraoperative visualization, thereby providing a safe, feasible, and cost-effective strategy for the surgical treatment of liver disease.

DETAILED DESCRIPTION:
The investigators have a series of surgical cases in which the investigators have been able to achieve excellent intraoperative biliary visualization with a greatly decreased (50-200 fold lower) dose of ICG than the previously published dose. Furthermore, this decreased dose was visible in about 15-20 minutes from the time of injection with low liver background fluorescence, a significant improvement that would make its utilization in the operating room more practical. The investigators hypothesize that a lower dose will: 1) allow adequate visualization of the extrahepatic biliary tree, including the cystic, common hepatic, and common bile ducts. Confirmation of hypotheses would mean that a lower dose of ICG can be administered on the same day of surgery in order to augment real-time intraoperative localization of the extrahepatic biliary tree, thereby providing a safe, feasible, and cost-effective strategy for the surgical treatment of liver disease.

The investigators intend to test our hypothesis with the following specific aims:

Aim 1: To compare the efficacy and utility of a low dose ICG (0.05 mg) protocol with a previously published dose (2.5 mg) in imaging the extrahepatic biliary tract.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing standard of care laparoscopic hepatic or biliary operations or Patients undergoing standard of care laparoscopic resection for hepatic tumors: hepatocellular carcinoma or metastatic tumor

Exclusion Criteria:

* Patients with a history of adverse reactions or known allergy to ICG, iodine, or iodine dyes and Pregnant and/or lactating patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zarrinpar, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Shands, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We are not sharing individual participant data with other researchers

REFERENCES:
- [Derived] Ladd AD, Zarate Rodriguez J, Lewis D, Warren C, Duarte S, Loftus TJ, Nassour I, Soma D, Hughes SJ, Hammill CW, Zarrinpar A. Low vs Standard-Dose Indocyanine Green in the Identification of Biliary Anatomy Using Near-Infrared Fluorescence Imaging: A Multicenter Randomized Controlled Trial. J Am Coll Surg. 2023 Apr 1;236(4):711-717. doi: 10.1097/XCS.0000000000000553. Epub 2023 Jan 10. PMID 36728303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing a planned laparoscopic cholecystectomy were approached between September 2021 to August 2022 in pre-surgical clinic and consented for a randomized ICG dose administration.
Pre-assignment Details: No enrolled patients were excluded from the study prior to group assignment.
Groups:
- Standard Dose: Prior to surgery these patients will be given a ICG dose of 2.5 mg IV.
  Indocyanine green: Low dose or standard dose ICG will be administered by the anesthesiologist as guided by the study coordinator at the beginning of the case, at two points during the operation (1- prior to the dissection of the biliary tract and 2- upon completion of the dissection and establishment of the critical view of safety).
Period: Overall Study
Arm/Group | Low Dose | Standard Dose
Started | 32 | 28
Completed | 32 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 5 enrolled and randomized patients were excluded from analysis because their videos were either too dark or unusable due to technical issues with the scope, camera, or device tower.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Standard Dose | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 20 | 46
  >=65 years | 6 | 8 | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [42 to 60] | 60 [42.3 to 65.8] | 57 [41.5 to 64.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  White | 26 | 24 | 46
  Black | 6 | 3 | 8
  Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Assessment - Bile Duct-to-liver Fluorescence Intensity Ratio
Description: Measurement is performed by dividing the fluorescence intensity signal of the common bile duct by that of the liver
Time Frame: intraoperative, average of 2 hours
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 29 | 26
ratio | 2.7 [1.5 to 4.2] | 0.7 [0.6 to 0.8]

2. Secondary Outcome: Qualitative Assessment of Overall Intraoperative Visualization of the Extrahepatic Biliary Tree - NIRFC Versus White Light
Description: A qualitative assessment will be made based on the quality of the intraoperative visualization of the extrahepatic biliary tree on a scale of 1 to 5 (1 = no improvement/identification not confirmed; 2 = marginally improved; 3 = sufficiently improved; 4 = well improved; 5 = greatly improved/exceeds expectations).
Time Frame: intraoperative, average of 2 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 29 | 26
score on a scale | 3.4 (1.3) | 3.1 (1.0)

3. Secondary Outcome: Quantitative Assessment - Bile Duct-to-background Fat Fluorescence Intensity Ratio
Description: Measurement is performed by dividing the fluorescence intensity signal of the common bile duct by that of the background fat
Time Frame: intraoperative, average of 2 hours
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 29 | 26
ratio | 6.1 [4.9 to 10.5] | 2.7 [2.4 to 3.0]

4. Secondary Outcome: Qualitative Assessment of Overall Intraoperative Visualization of the Extrahepatic Biliary Tree (Common Hepatic Duct, Cystic Duct, Common Bile Duct, Aberrant Ducts)
Description: as for outcome 2
Time Frame: intraoperative, average of 2 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 29 | 26
score on a scale
  Common Hepatic Duct | 3.6 (1.4) | 2.8 (1.3)
  Cystic Duct | 3.6 (1.3) | 3.5 (1.2)
  Common Bile Duct | 3.6 (1.3) | 3.1 (1.3)
  Aberrant Duct | 2.8 (1.3) | 2.3 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, an average of 24 hours.
Description: ICG is a very safe drug with minimal risk for adverse advents. Participants were given a very low dose
Groups:
- Low Dose: Study participants who received low dose ICG.
- Standard Dose: Study participants who received standard dose ICG.
Arm/Group | Low Dose | Standard Dose
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26
Other Adverse Events (participants affected / at risk) | 0/29 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04942665/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04942665/SAP_001.pdf
  • Informed Consent Form (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT04942665/ICF_002.pdf